CLINICAL TRIAL: NCT05349500
Title: Optimizing Osteoarthritis Care Through Clinical and Community Partnership
Brief Title: OA Clinic-Community CARE Model
Acronym: OA CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0865; 1R21AR080309-01 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Overweight; Obesity; Physical Inactivity; Weight Loss
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Overweight; Obesity; Sedentary Behavior; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA CARE (Experimental): Participants assigned to the OA CARE intervention will receive a 12-month Medical Membership to a local YMCA and participate in a 12-week weight loss program. Participants will also work with an OA CARE Navigator, who, in partnership with their primary care provider (PCP), will identify any additional programs or resources that may help them manage their osteoarthritis (OA) symptoms.
  Interventions: Behavioral: OA CARE Intervention
- Usual Care (Placebo Comparator): Participants assigned to this group will receive no additional treatment from the study for about 12 months.
  Interventions: Behavioral: Usual Care control group

INTERVENTIONS:
Behavioral: OA CARE Intervention — Once assigned, participants will be contacted by the OA CARE Navigator to coordinate initiating a YMCA Medical Membership. Then, YMCA personnel will contact the participant to schedule the first Weight Loss Program (Program) group session. The Program will be delivered in groups with other OA CARE participants. Participants will also have access to all exercise facilities and programs at the YMCA during the study, and will be assigned a YMCA health coach.
  After initiation of the YMCA Medical Membership, the OA CARE Navigator will discuss participant's interests in referrals to other services related to osteoarthritis (OA) management. The Navigator will provide the participant's primary care provider (PCP) with a summary of this discussion and help the participant connect to any programs or resources that do not require provider referrals.
  Arms: OA CARE
Behavioral: Usual Care control group — Participants assigned to the usual care group will receive no additional treatment from the study for about 12 months. However, this group will be offered a 12-month Medical Membership to a local YMCA after completing the final assessment.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to test the OA Clinic-Community CARE Model (OA CARE) which will address all recommended components of knee/hip (osteoarthritis) OA care, include interventions for both patients and primary care providers (PCPs), and utilize a tailored approach that efficiently matches treatments with patients' needs.

The patient component of OA CARE will include evidence-based weight management and exercise programs for all participants (delivered through the YMCA), as well as tailored referrals to physical therapy, additional weight management or nutrition services, sleep-related services and psychological services.

The PCP component of OA CARE will include a video-based summary of current OA treatment guidelines (with emphasis on practical application), collaboration on patients' referrals to specific services described above, and progress reports on enrolled patients.

DETAILED DESCRIPTION:
This study will be a randomized pilot trial of OA CARE among n=60 patients with knee and/or hip osteoarthritis (OA) and overweight/obesity who are not currently meeting physical activity recommendations. Participants will be randomly assigned to OA CARE or a usual care (UC) group. Assessments will be conducted at baseline, 6 months and 12 months. Primary endpoint of the trial will be self-reported pain and function and secondary endpoint will be objectively assessed physical activity (PA), measured via accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of knee or hip OA
* Self-reported knee or hip pain of ≥3 (scale of 0-10) on most days of the week
* Current Weekly Physical Activity <150 minutes per week
* Body mass index (BMI) ≥27 kg/m^2

Exclusion Criteria:

* No internet access and a device (computer, tablet, smartphone) to access the virtual weight loss intervention
* Pain in chest when performing physical activity
* Pain in chest when not performing physical activity
* No documented diagnosis of knee or hip OA
* Total knee or hip replacement surgery, meniscus tear, ligament tear, or other significant lower extremity injury or surgery in the last 6 months
* Dementia or other memory loss condition
* Active diagnosis of psychosis
* Active Substance abuse disorder
* Severe hearing or visual impairment
* Serious/terminal illness as indicated by referral to hospice or palliative care
* Hospitalization for cardiovascular event in last 6 months
* History of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (2 hospitalizations within the previous 6 months and/or on oxygen)
* Stroke with moderate to severe aphasia
* Recent history (last 6 months) of three or more falls
* Planning total joint replacement in next 6 months
* Any other health conditions determined by the study team to be contraindications to a home exercise program or weight loss
* Current participation in other study related to knee or hip osteoarthritis or physical activity
* Unable to speak English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/ sharing agreement with University of North Carolina at Chapel Hill (UNC).
Supporting Information: SAP
Time Frame: Data will become available following publication of primary and secondary outcomes. Research study records will be maintained for no less than 6 years following the completion of the study.
Access Criteria: Data will be accessible following publication of study results and will be available for no less than 6 years following the completion of the study.

RESULTS

PARTICIPANT FLOW:
Groups:
- OA CARE: Participants assigned to the OA CARE intervention will receive a 12-month Medical Membership to a local YMCA and participate in a 12-week weight loss program. Participants will also work with an OA CARE Navigator, who, in partnership with their primary care provider (PCP), will identify any additional programs or resources that may help them manage their osteoarthritis (OA) symptoms.
  OA CARE Intervention: Once assigned, participants will be contacted by the OA CARE Navigator to coordinate initiating a YMCA Medical Membership. Then, YMCA personnel will contact the participant to schedule the first Weight Loss Program (Program) group session. The Program will be delivered in groups with other OA CARE participants. Participants will also have access to all exercise facilities and programs at the YMCA during the study, and will be assigned a YMCA health coach.
  After initiation of the YMCA Medical Membership, the OA CARE Navigator will discuss participant's interests in referrals to other services related to osteoarthritis (OA) management. The Navigator will provide the participant's primary care provider (PCP) with a summary of this discussion and help the participant connect to any programs or resources that do not require provider referrals.
Period: Overall Study
Arm/Group | OA CARE | Usual Care
Started | 30 | 30
Completed | 23 | 24
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OA CARE | Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.5) | 65.6 (9.1) | 64.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 17 | 20 | 37
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
WOMAC Total Score [Mean (Standard Deviation); unit: units on a scale] — For the WOMAC total score, the test questions are scored on a scale of 0-4. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The overall WOMAC score is determined by summing the scores for all three subscales and the score ranges include 0-96 (derived from a 0-4 Likert scale), with higher scores indicating worse pain, stiffness, and functional limitations.
  units on a scale | 40.7 (14.4) | 37.9 (17.3) | 39.3 (15.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 6 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Total Score
Description: For the WOMAC total score, the test questions are scored on a scale of 0-4. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The overall WOMAC score is determined by summing the scores for all three subscales and the score ranges include 0-96 (derived from a 0-4 Likert scale), with higher scores indicating worse pain, stiffness, and functional limitations.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed both baseline and 6-month follow-up assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 24 | 27
units on a scale | -7.8 [-16.04 to 0.4] | 3.2 [-4.8 to 11.2]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-20.1 to -1.9]

2. Primary Outcome: Change From Baseline to Month 12 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Total Score
Description: as for outcome 1
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month follow-up assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 23 | 24
units on a scale | -8.3 [-16.4 to -0.2] | -3.3 [-11.3 to 4.6]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.286, Mixed Models Analysis; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-14.1 to 4.3]

3. Secondary Outcome: Change From Baseline to Month 6 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: The WOMAC Pain Subscale is a measure of lower extremity pain. It includes 5 items rated on a Likert scale of 0 (no pain) to 4 (extreme pain), with a total range of 0-20 with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed baseline and 6-month follow-up assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 24 | 27
units on a scale | -1.5 [-3.6 to 0.5] | 0.5 [-1.6 to 2.5]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.0 to -0.0]

4. Secondary Outcome: Change From Baseline to Month 12 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: as for outcome 3
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed baseline and 12-month follow-up assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 23 | 24
units on a scale | -2.1 [-4.1 to -0.0] | -0.4 [-2.5 to 1.6]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.8 to 0.5]

5. Secondary Outcome: Change From Baseline to Month 6 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: The WOMAC function subscale includes 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty), with ranges of 0-68 for the function subscale with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed baseline and 6-month follow-up assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 24 | 27
units on a scale | -4.9 [-10.6 to 0.7] | 2.6 [-2.8 to 8.0]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.031, Mixed Models Analysis; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-14.3 to -0.7]

6. Secondary Outcome: Change From Baseline to Month 12 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: as for outcome 5
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed baseline and 12-month follow-up assessments
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 23 | 24
units on a scale | -4.5 [-10.1 to 1.0] | -2.6 [-7.9 to 2.8]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.564, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-8.8 to 4.9]

7. Secondary Outcome: Change From Baseline to Month 6 in Objectively Assessed Physical Activity Per Week (Accelerometer), Log Transformed.
Description: Minutes of moderate to vigorous intensity physical activity (MVPA) per week measured via accelerometer.
  This measure was log transformed because raw data did not meet assumptoms for statsitical models.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed baseline and 6-month accelerometer assessments. Note that some participants completed follow-up questionnaires but not accelerometer wear.
Measure: Mean (95% Confidence Interval); unit: log (minutes / week)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 22 | 25
log (minutes / week) | 0.2 [-0.2 to 0.5] | -0.0 [-0.3 to 0.3]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.349, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]

8. Secondary Outcome: Change From Baseline to Month 12 in Objectively Assessed Physical Activity Per Week (Accelerometer), Log Transformed
Description: as for outcome 7
Time Frame: Baseline, Month 12 (Follow-up)
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: log (minutes / week)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 20 | 20
log (minutes / week) | -0.3 [-0.6 to 0.1] | -0.1 [-0.4 to 0.3]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.303, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.2]

9. Secondary Outcome: Change From Baseline to Month 6 in Steps Per Day, Log Transformed
Description: Step counts measured via accelerometer. This measure was log transformed because raw data did not meet assumptoms for statsitical models.
Time Frame: Baseline, Month 6 (Follow-up)
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: log (steps / day)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 22 | 25
log (steps / day) | 0.00 [-0.2 to 0.3] | -0.0 [-0.3 to 0.2]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.507, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.1 to 0.2]

10. Secondary Outcome: Change From Baseline to Month 12 in Steps Per Day, Log Transformed
Description: as for outcome 9
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed baseline and 12-month accelerometer assessments. Note that some participants completed follow-up questionnaires but not accelerometer wear.
Measure: Mean (95% Confidence Interval); unit: log (steps / day)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 20 | 20
log (steps / day) | -0.1 [-0.3 to 0.2] | -0.1 [-0.4 to 0.1]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.729, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

11. Secondary Outcome: Change From Baseline to Month 6 in Minutes of Any Physical Activity (PA) Per Day, Standardized to a 16 Hour Day
Description: Minutes of any PA measured via accelerometer. This measure was standardized to a 16 hour day to address between-patient differences in amount of wear time.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed both baseline and 6-month follow-up acceleromter assessments. Note that some participants completed questionnaires but not accelerometer wear.
Measure: Mean (95% Confidence Interval); unit: minutes / day
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 22 | 25
minutes / day | -0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.421, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

12. Secondary Outcome: Change From Baseline to Month 12 in Minutes of Any Physical Activity (PA) Per Day, Standardized to 16 Hour Day
Description: as for outcome 11
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month follow-up acceleromter assessments. Note that some participants completed questionnaires but not accelerometer wear.
Measure: Mean (95% Confidence Interval); unit: min/day
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 20 | 20
min/day | -0.1 [-0.2 to 0.0] | -0.1 [-0.2 to 0.1]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.648, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.2 to 0.1]

13. Secondary Outcome: Change From Baseline to Month 6 in Self-Reported Minutes of Moderate to Vigorous Physical Activity Per Week, Square Root Transformed
Description: Self-Reported Physical Activity will be assessed using the Modified version of the CHAMPS (Community Health Activities Model Program for Seniors) Physical Activity Measure. Data from the questionnaire is used to determine variety, frequency, and minutes per week from physical activity. Separate scores are derived for physical activities of moderate or greater intensity (metabolic equivalents MET ≥ 3.0) and for all activities listed (light, moderate, and vigorous). Estimates of frequency (days per week) range from 0 to 7 days per week. Estimates of Variety (# different activities), while open, generally ranges from 0 to 5, values above 5 are checked. Estimates of minutes, generally range from 0 to 180 per day. Individuals reporting more than 180 minutes per day are checked. For all physical activity outcomes higher values equal a greater amount of activity. This measure was square root transformed becuase raw failed to meet assumptions for statistical analyses.
Time Frame: Baseline, Month 6 (Follow-up)
Population: Participants who completed baseline and 6-month questionnaires
Measure: Mean (95% Confidence Interval); unit: square root (minutes per week)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 24 | 27
square root (minutes per week) | 4.6 [2.3 to 6.9] | 1.2 [-0.9 to 3.3]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.034, Mixed Models Analysis; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [0.3 to 6.5]

14. Secondary Outcome: Change From Baseline to Month 12 in Self-Reported Minutes of Moderate to Vigorous Physical Activity Per Week, Square Root Transformed
Description: Self-Reported Physical Activity will be assessed using the Modified version of the CHAMPS (Community Health Activities Model Program for Seniors) Physical Activity Measure. Data from the questionnaire is used to determine variety, frequency, and minutes per week from physical activity. Separate scores are derived for physical activities of moderate or greater intensity (metabolic equivalents (MET) ≥ 3.0) and for all activities listed (light, moderate, and vigorous). Estimates of frequency (days per week) range from 0 to 7 days per week. Estimates of Variety (# different activities), while open, generally ranges from 0 to 5, values above 5 are checked. Estimates of minutes, generally range from 0 to 180 per day. Individuals reporting more than 180 minutes per day are checked. For all physical activity outcomes higher values equal a greater amount of activity.
  This measure was square root transformed because raw data did not meet assumptions for statistical models.
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed baseline and 12-month questionnaires
Measure: Mean (95% Confidence Interval); unit: square root (minutes per week)
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 23 | 24
square root (minutes per week) | 4.3 [1.3 to 7.3] | 2.2 [-0.7 to 5.1]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.315, Mixed Models Analysis; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-2.1 to 6.3]

15. Secondary Outcome: Change From Baseline to Month 6 in Sedentary Minutes Per Day, Standardized to a 16 Hour Day
Description: Sedentary minutes measured via accelerometer This measure was standardized to a 16 hour day to address between-patient differences in amount of wear time.
Time Frame: Baseline, Month 6 (Follow-up)
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: minutes / day
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 22 | 25
minutes / day | 10.5 [-15.1 to 36.1] | -2.9 [-26.4 to 20.6]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.444, Mixed Models Analysis; Mean Difference (Final Values) = 13.4, 95% CI 2-sided [-21.5 to 48.2]

16. Secondary Outcome: Change From Baseline to Month 12 in Sedentary Minutes Per Day, Standardized to a 16 Hour Day
Description: as for outcome 15
Time Frame: Baseline, Month 12 (Follow-up)
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: minutes / day
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 20 | 20
minutes / day | 18.6 [-9.6 to 46.9] | 9.3 [-18.6 to 37.2]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.638, Mixed Models Analysis; Mean Difference (Final Values) = 9.3, 95% CI 2-sided [-30.6 to 49.2]

17. Secondary Outcome: Change From Baseline to Month 12 in Body Weight
Description: Body weight assessed using a research / clinical grade scale (e.g., Tanita) that will be calibrated regularly.
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month follow-up weight assessment.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 23 | 22
kg | -7.6 [-15.5 to 0.4] | -5.4 [-13.0 to 2.3]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.688, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-13.4 to 8.9]

18. Secondary Outcome: Change From Baseline to Month 12 in 30-second Chair Stand Test
Description: Assessed to test participant leg strength and endurance. Measured by total number of chair stands (up and down equals one stand) completed in 30 seconds.
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month follow-up chair stand tests.
Measure: Mean (95% Confidence Interval); unit: number of chair stands in 30 seconds
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 14 | 21
number of chair stands in 30 seconds | -0.9 [-2.5 to 0.7] | -0.6 [-1.8 to 0.7]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.709, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.5 to 1.7]

19. Secondary Outcome: Change From Baseline to Month 12 in Timed Up-and-go (TUG) Test
Description: Assessed to measure participant functional mobility. Measured by how many seconds it takes for participant to stand up, walk to the mark, turn around, return & sit back into a chair with their back resting on the back of the chair.
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month TUG tests.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 15 | 12
seconds | 0.5 [-0.9 to 1.8] | 2.0 [0.9 to 3.1]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.089, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.3 to 0.2]

20. Secondary Outcome: Change From Baseline to Month 12 in 2-minute March Test
Description: Assessed to evaluate participant functional aerobic endurance. Measured by number of steps completed in 2 minutes.
Time Frame: Baseline, Month 12 (Follow-up)
Population: Participants who completed both baseline and 12-month follow-up 2-minute march tests.
Measure: Mean (95% Confidence Interval); unit: steps
Arm/Group | OA CARE | Usual Care
Number analyzed (Participants) | 14 | 21
steps | 29.7 [17.4 to 42.0] | 14.8 [4.9 to 24.7]
Statistical Analysis 1: Comparison: OA CARE vs Usual Care; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = 14.9, 95% CI 2-sided [-1.0 to 30.8]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | OA CARE | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT05349500/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT05349500/ICF_000.pdf